CLINICAL TRIAL: NCT03102307
Title: A Prospective, Multicenter, Registry Trial to Evaluate Utilization Frequency and Feasibility of Targeted Axillary Dissection (TAD) After Needle Biopsy and Clip Placement in Early Breast Cancer With Clinically Affected Lymph Nodes
Brief Title: Registry Trial to Evaluate the Clinical Utilization of Targeted Axillary Dissection (TAD)
Status: Completed | Type: Observational
Sponsor: Kliniken Essen-Mitte (Other)
Collaborators: GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: SenTa
Record Dates: First submitted 2017-03-27; First posted 2017-04-05 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Early Stage Breast Cancer
Keywords: Targeted axillary dissection; Sentinel node biopsy; Neoadjuvant chemotherapy
MeSH Terms: interventions — DAT protocol 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CNB biopsy/clip placement not done: Clinically affected lymph nodes cannot be biopsied or clip labeled. Patients are not suitable for TAD
  Interventions: Other: Not suitable for TAD
- CNB/clip placement done - benign: Clinically affected lymph nodes can be biopsied and clip labeled. Needle biopsy reveals no axillary tumor spread. Patients are suitable for TAD
  Interventions: Procedure: Suitable for TAD
- CNB/clip placement done - malignant: Clinically affected lymph nodes can be biopsied and clip labeled. Needle biopsy reveals axillary tumor spread. Patients are suitable for TAD
  Interventions: Procedure: Suitable for TAD

INTERVENTIONS:
Other: Not suitable for TAD — Registry of the rate of patients not suitable for TAD as initial CNB with clip placement of axillary lymph nodes is not possible and underlying medical contraindications, technical obstacles or miscellaneous reasons why needle biopsy and/or clip labeling of clinically affected lymph nodes cannot be done
  Groups: CNB biopsy/clip placement not done
Procedure: Suitable for TAD — Registry of surgical outcome measures of targeted resection of the clipped node with optional sentinel node biopsy or axillary lymph node dissection with or without preceding neoadjuvant chemotherapy
  Groups: CNB/clip placement done - benign; CNB/clip placement done - malignant

SUMMARY:
A downstaging of axillary tumor-spread can be achieved in about 40% of the patients receiving neoadjuvant chemotherapy (NACT). The impact of NACT on loco-regional tumor control has not yet been sufficiently investigated. Moreover the pathologic nodal status after NACT is a strong prognostic marker. Therefore it is most desirable to identify the approximately 40% of patients with pathologic complete response of the axilla, that could be spared from a potentially non beneficial axillary lymph node dissection (ALND). Attempts to identify these patients via sentinel lymph node biopsy (SLNB) after NACT have failed to provide acceptable false negative rates (FNR). The new concept of targeted axillary dissection (TAD) following NACT has shown promising results. Still multiple information about the clinical adoption of this procedure into clinical practice are missing. The SenTa registry trial is designed to assess the clinical implementation of TAD into general practice.

DETAILED DESCRIPTION:
For decades the pathologic nodal status in early breast cancer has been of paramount importance, when evaluating the need for further adjuvant therapies. Nowadays tumor characteristics as receptor status and gene expression essays are increasingly included in this decision process. An increasing number of breast cancer patients are treated with neoadjuvant chemotherapy (NACT). A downstaging of axillary tumor-spread can be achieved in about 40% of the patients receiving NACT. The contribution of NACT to loco-regional tumor control is not fully integrated into the surgical treatment plan. The introduction of sentinel lymph node biopsy (SLNB) and the results of the ACOSOG (American College of Surgeons Oncology Group) Z0011 trial led to a reduction in radicalness of axillary surgery in the adjuvant setting. The impact of NACT on loco-regional tumor control in the neoadjuvant setting has not yet been sufficiently investigated. Moreover the pathologic nodal status after NACT is a strong prognostic marker. Therefore it is most desirable to identify the approximately 40% of patients with pathologic complete response of the axilla and distinguish these patients from those with tumor residuals which might need additional postneoadjuvant treatment. So far attempts to identify these patients via SLNB after NACT have failed to provide acceptable false negative rates (FNR) as reported in the SENTINA (Sentinel-lymph-node biopsy in patients with breast cancer before and after neoadjuvant chemotherapy) trial and ACOSOG Z1071 trial.

Attempts have bee made to further improve FNR of SLNB after NACT in patients with clinically affected lymph nodes at initial presentation. A new concept of surgical axillary staging after NACT is the targeted axillary dissection (TAD). First results have shown to reduce FNR far below the desired threshold of 10%. In this procedure clinically suspicious lymph nodes are evaluated by core needle biopsy (CNB) or fine needle aspiration (FNA) before NACT. A clip is placed into the most suspicious appearing lymph node (target lymph node TLN) directly after biopsy. In case of proven metastasis surgical staging of the axilla is postponed to after completion of NACT. The targeted resection of the clipped node after NACT (target lymph node biopsy TLNB) displays a FNR of 2 - 4.2% according to first results published by Caudle et al. in 2016. In about 3 out of 4 patients the TLN equals a SLN if SLNB is performed simultaneously. The combination of TLNB and SLNB (together so called TAD) seems to further lower FNR. Cases in which tracer uptake in lymph nodes is impaired i.e. by tumor residuals and presumably result in a false negative SLNB can be covered by TLNB.

Clip placement in affected axillary lymph nodes for the purpose of following targeted resection has been implemented into international guidelines. But to date multiple insights into clinical application of TAD are missing. It is not known how often initial CNB/FNA of axillary lymph nodes and following clip placement is successful or has to be abandoned because of technical/medical contraindications. Moreover it is not known how often visualization of the clip after normalization of lymph node structures following NACT and month after initial clip placement is possible. Furthermore information about optimal clip material are lacking. In summary success rates for the targeted resection of the clipped node have to be investigated. Therefore the intraoperative detection rate of the clipped target lymph node is our primary outcome measure.

Patients with clinically affected lymph nodes at initial presentation are planned to be enrolled in multiple german breast centers. In accorndance to german guidelines it is aimed to evaluate the pathologic nodal status via CNB with following clip placement in all of these patients after informed consent. If CNB or clip placement cannot be achieved, technical/medical contraindications are recorded. As the SenTa trial is a registry trial, no strict directives for the further surgical treatment are made. If clip placement is successful, further procedures are left at the investigators choice according to initial pathologic nodal status and potential clinical response to NACT.

If no tumor manifestations are detected in initial CNB, SLNB with simultaneous targeted resection of the clipped node (TLNB) is recommended. The rationale for TLNB in this situation is a FNR of about 20% of initial CNB. On an individual basis upfront ALND can be offered.

If tumor manifestations are detected in initial CNB, targeted resection of the clipped node (TLNB) is strongly recommended because of obvious reasons. If NACT is not planned, upfront ALND should be offered. If patients are planned for NACT further procedures are left at the investigators discretion according to clinical response to NACT. Clinical response after NACT is assessed by axillary ultrasound and an optional needle biopsy if applicable. In case of clinical complete response, TLNB with simultaneous SLNB can be offered on an individual basis.

ELIGIBILITY:
Inclusion Criteria

* informed consent
* invasive mamma carcinoma verified by needle biopsy of the primary tumor
* nodal positive (cN+) verified by axillary ultrasound
* cT stage 1-4c, multifocality allowed
* no sign of distant metastasis (cM0)

Exclusion Criteria:

* prior history of breast cancer
* prior ipsilateral extensive surgery of breast or axilla
* inflammatory or extramammary breast cancer
* pregnancy
* inability to understand the studies purpose
* no written patient informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed invasive breast cancer with clinically affected lymph nodes
Sampling Method: Non-Probability Sample
Enrollment: 548 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Surgical detection rate of the clip labeled target lymph node | 6 month for patients undergoing NACT after initial needle biopsy/clip placement and subsequent surgical resection of the clipped node
  Successful intraoperative detection and targeted resection of clip labeled target lymph node as confirmed by specimen radiography and/or surgeon

SECONDARY OUTCOMES:
Rate of patients not suitable for targeted axillary dissection (TAD) | 14 days
  Rate of patients not suitable for TAD as initial CNB with clip placement of axillary lymph nodes is not possible and underlying medical contraindications, technical obstacles or miscellaneous reasons why needle biopsy and/or clip labeling of clinically affected lymph nodes cannot be done
Rate of representative and successful lymph node CNB | 14 days
  Rate of CNB revealing tumor manifestations or lymph node tissue on histology out of all performed lymph node CNB
Rate of preoperative sonographic clip detection | 6 month for patients undergoing NACT after initial needle biopsy/clip placement and subsequent surgical resection of the clipped node
  Essential requirement for targeted resection of the clipped target lymph node is the preoperative visualization of the clip for the purpose of guide wire localization
Rate of patients treated with TAD after NACT | 6 month for patients undergoing NACT after initial needle biopsy/clip placement and subsequent surgical resection of the clipped node
  Rate of patients with intraoperative detection of at least one sentinel lymph node and the clip labeled target lymph node as confirmed by specimen radiography and/or surgeon
Rate of patients treated with upfront ALND after NACT | 6 month for patients undergoing NACT after initial needle biopsy/clip placement and subsequent surgical resection of the clipped node
  Rate of patients treated with upfront axillary dissection including resection of clipped node after completion of NACT
False negative rate for target lymph node biopsy (TLNB) alone | 6 month for patients undergoing NACT after initial needle biopsy/clip placement and subsequent surgical resection of the clipped node
  Clipped target lymph node does not contain tumor manifestations after NACT but lymph node metastasis is revealed by ALND
False negative rate for Sentinel Lymph Node Biopsy (SLN) alone | 6 month for patients undergoing NACT after initial needle biopsy/clip placement and subsequent surgical resection of the clipped node
  Sentinel lymph node does not contain tumor manifestations after NACT but lymph node metastasis is revealed by ALND
Detection Rate for Targeted Axillary Detection (TAD) (SLN and TLN detected) | 6 month for patients undergoing NACT after initial needle biopsy/clip placement and subsequent surgical resection of the clipped node
  Successful intraoperative detection and resection of at least one sentinel lymph node and the clip labeled target lymph node as confirmed by specimen radiography and/or surgeon
Detection Rate for Sentinel Lymph Node Biopsy (SLNB) | 6 month for patients undergoing NACT after initial needle biopsy/clip placement and subsequent surgical resection of the clipped node
  Successful intraoperative detection and resection of at least one sentinel lymph node
Rate of patients,where the clip is found in a sentinel lymph node (SLN) | 6 month for patients undergoing NACT after initial needle biopsy/clip placement and subsequent surgical resection of the clipped node
  Clip is located in a sentinel lymph node during TAD, hence the TLN equals a SLN
Number of excised lymph nodes during targeted axillary dissection (TAD) | 6 month for patients undergoing NACT after initial needle biopsy/clip placement and subsequent surgical resection of the clipped node
  Number of excised lymph nodes during targeted axillary dissection (TAD) equals count of sentinel lymph nodes plus target lymph nodes
Number of excised lymph nodes during sentinel lymph node biopsy (SLNB) | 6 month for patients undergoing NACT after initial needle biopsy/clip placement and subsequent surgical resection of the clipped node
  Number of excised lymph nodes during targeted axillary dissection (TAD) equals count of sentinel lymph nodes plus target lymph nodes
Number of excised target lymph nodes (TLN) which are not a sentinel lymph node | 6 month for patients undergoing NACT after initial needle biopsy/clip placement and subsequent surgical resection of the clipped node
  Number of excised clipped lymph nodes during target lymph node biopsy (TLNB) which are not sentinel lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: Sherko Kümmel, MD, Principal Investigator — Kliniken Essen-Mitte; Johannes Holtschmidt, MD, Study Chair — Kliniken Essen-Mitte; Thortsen Kühn, MD, Study Chair — Klinikum Esslingen
Locations (3):
- Germany (3):
  - Kliniken Essen-Mitte, Essen, North Rhine-Westphalia
  - Klinikum Esslingen, Esslingen am Neckar
  - Evangelische Kliniken Gelsenkirchen, Gelsenkirchen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caudle AS, Yang WT, Krishnamurthy S, Mittendorf EA, Black DM, Gilcrease MZ, Bedrosian I, Hobbs BP, DeSnyder SM, Hwang RF, Adrada BE, Shaitelman SF, Chavez-MacGregor M, Smith BD, Candelaria RP, Babiera GV, Dogan BE, Santiago L, Hunt KK, Kuerer HM. Improved Axillary Evaluation Following Neoadjuvant Therapy for Patients With Node-Positive Breast Cancer Using Selective Evaluation of Clipped Nodes: Implementation of Targeted Axillary Dissection. J Clin Oncol. 2016 Apr 1;34(10):1072-8. doi: 10.1200/JCO.2015.64.0094. Epub 2016 Jan 25. PMID 26811528
- [Background] Boughey JC, Suman VJ, Mittendorf EA, Ahrendt GM, Wilke LG, Taback B, Leitch AM, Kuerer HM, Bowling M, Flippo-Morton TS, Byrd DR, Ollila DW, Julian TB, McLaughlin SA, McCall L, Symmans WF, Le-Petross HT, Haffty BG, Buchholz TA, Nelson H, Hunt KK; Alliance for Clinical Trials in Oncology. Sentinel lymph node surgery after neoadjuvant chemotherapy in patients with node-positive breast cancer: the ACOSOG Z1071 (Alliance) clinical trial. JAMA. 2013 Oct 9;310(14):1455-61. doi: 10.1001/jama.2013.278932. PMID 24101169
- [Background] Kuehn T, Bauerfeind I, Fehm T, Fleige B, Hausschild M, Helms G, Lebeau A, Liedtke C, von Minckwitz G, Nekljudova V, Schmatloch S, Schrenk P, Staebler A, Untch M. Sentinel-lymph-node biopsy in patients with breast cancer before and after neoadjuvant chemotherapy (SENTINA): a prospective, multicentre cohort study. Lancet Oncol. 2013 Jun;14(7):609-18. doi: 10.1016/S1470-2045(13)70166-9. Epub 2013 May 15. PMID 23683750
- [Result] Kuemmel S, Heil J, Rueland A, Seiberling C, Harrach H, Schindowski D, Lubitz J, Hellerhoff K, Ankel C, Grasshoff ST, Deuschle P, Hanf V, Belke K, Dall P, Dorn J, Kaltenecker G, Kuehn T, Beckmann U, Potenberg J, Blohmer JU, Kostara A, Breit E, Holtschmidt J, Traut E, Reinisch M. A Prospective, Multicenter Registry Study to Evaluate the Clinical Feasibility of Targeted Axillary Dissection (TAD) in Node-positive Breast Cancer Patients. Ann Surg. 2022 Nov 1;276(5):e553-e562. doi: 10.1097/SLA.0000000000004572. Epub 2020 Nov 4. PMID 33156057